CLINICAL TRIAL: NCT04457583
Title: Inspiratory Muscle Training on Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE49197915.3.0000.5256
Record Dates: First submitted 2018-08-16; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Inspiratory Muscle Training; Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Inspiratory Muscle Training; Life of quality
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Controlled and randomized clinical trial involving 70 patients with OSAHS diagnosed by polysomnography. Measurements of maximal inspiratory pressure (MIP) will be performed. Pittsburgh scale Epworth, Sleepiness Scale, Short Form-36, and Berlin / Stanford questionnaires will be used for assessment of sleep quality, daytime sleepiness, health related quality of life quality of health (QOL), and the evaluation of snoring. Patients of the intervention group will undergo IMT with an initial load of 40% of MIP. The intervention will be performed daily for 12 weeks employing the exercise inspiratory device (POWERbreathe, HaB Ltd, UK). The main end point will be the effect of the training program on the index of apnea / hypopnea (IAH) assessed by polysomnography. Secondary end points will include effects of the training program on: the quality of sleep, inspiratory muscle strength, the health related QOL
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Procedure: Inspiratory muscle training with powerbreathe with a linear pressure resistance using an inspiratory load of 40% of maximal inspiratory pressure (adjusted weekly), seven days a week, 30 exercises daily for 12 weeks.
  Interventions: Device: Inspiratory muscle training with powerbreathe
- Control (No Intervention): Procedure: Training with the same equipment but without load-generating resistance.

INTERVENTIONS:
Device: Inspiratory muscle training with powerbreathe — Participants will be submitted to a linear pressure resistance (Powerbreathe) with an inspiratory load of 40% of maximal inspiratory pressure (adjusted weekly), seven days a week, session duration of 30 exercises for 12 weeks.
  Arms: Intervention

SUMMARY:
Introduction: Studies have shown the influence of exercise on sleep architecture and efficiency, although its protocols, procedures, effects and mechanisms of action have not been clearly explained and documented in the treatment of obstructive sleep apnea hypopnea syndrome (OSAHS), which is thought to be the main sleep disorder due to its high prevalence and clinical, social and cognitive consequences. Objective: To evaluate the effect of inspiratory muscle training (IMT) in OSAHS, by analyzing their influence on the quality of sleep, inspiratory muscle strength and polysomnography parameters. Patients and Methods: Controlled and randomized clinical trial involving 75 patients with OSAHS diagnosed by polysomnography. Measurements of maximal inspiratory pressure (MIP) will be performed. Pittsburgh scale Epworth, Sleepiness Scale, Short Form-36, and Berlin / Stanford questionnaires will be used for assessment of sleep quality, daytime sleepiness, health related quality of life quality of health, and the evaluation of snoring. Patients of the intervention group will undergo IMT with an initial load of 40% of MIP. The intervention will be performed daily for 12 weeks employing the exercise inspiratory device (POWERbreathe, HaB Ltd, UK). The main end point will be the effect of the training program on the index of apnea/hypopnea (IAH) assessed by polysomnography. Secondary end points will include effects of the training program on: the quality of sleep, inspiratory muscle strength, the health related QOL. Expected Results: if the hypothesis is confirmed, there will be improvements on the apnea / hypopnea index, on the quality of sleep and on the health related QOL.

DETAILED DESCRIPTION:
MATERIAL AND METHODS Study population Studied population will be derived from the Hospital Naval Marcilio Dias (HNMD), the sample consisting of active military personnel, reserve personnel and members of the naval family who seek the otorhinolaryngology service of the hospital.

Participants will be instructed about the objectives and methods of the present study and, in order to participate in the study, will be consulted to give their written consent for inclusion, according to the Informed Consent Term.

Study Design Study will be conducted through a prospective, controlled, randomized, and masked clinical trial for the participants and the investigator who will perform the data analysis.

Sample Characterization Reference Population It will consist of patients in medical care at the otorhinolaryngology clinic of Naval Hospital Marcílio Dias (HNMS), referred for polysomnography with a view to diagnosing OSAHS, obeying inclusion and exclusion criteria. All patients referred will be receiving the standard treatment for OSAHS, which consists of the nocturnal use of CPAP.

The stratified random probabilistic sample will consist of 2 (two) groups, control (sham) and intervention. Participants will be consecutively allocated in the intervention or control group by order of entry into the study and by level of severity of OSAHS to ensure fairness between groups regarding OSAHS severity.

Sample size The sample size was estimated through calculations to be able to evaluate differences of the order of 20% between the groups, with a power of 80% and an alpha error of 5%, with a quantitative of 35 patients per group, totaling 70 (Seventy) patients.

Characterization of groups and IMT protocol All patients will receive standard medical treatment, which usually includes use of nocturnal CPAP. The intervention group will receive inspiratory muscle training, through 30 respiratory cycles in the POWERbreathe classic, with an initial load of 40% of PImax, once a day, during the 7 days of the week, for 02 weeks. An increase of 01 level in the resistance of the POWERbreathe classic, equivalent to an increase of 10 cmH2O, will be carried out at the beginning of the third, fourth and fifth weeks.

From the sixth to twelfth week, the resistance will not be increased further, remaining at the value of the last adjustment. The sham control group will be submitted to exercises with the same apparatus, but without load. The IMT program will begin with a (01) supervised care, in which the research protocol will be presented to the patient, explaining the steps of the research, when supervised orientation of the IMT will be performed and awareness about the importance of adherence to the treatment. If the patient persists, before starting the research protocol, the patient will be heard and given the pertinent guidelines until all their doubts are resolved so that they can be selected for the intervention group.

In the initial stage of the protocol, the patient will receive guidance containing information to assist in the correct implementation of the MRI and a record sheet of daily MRI achievement, allowing uniformity and documentation of its achievement, respectively.

At the end of every 04 weeks, patients will attend the HNMD physical therapy service for follow-up and clinical reassessment. At the end of 12 weeks, they will attend the last clinical and polysomnographic evaluation. Throughout the period the patients in the study will be performing IMT.

To promote adherence to research, patients will receive guidance on how the equipment works, how it is used, frequency and duration of exercise; As well as follow-up through scheduled appointments. Phone calls will be made bi-weekly to certify that protocols, motivational messages, follow-up phone calls and confirmation of appointments marked for protocol reassessment are still in progress.

Instrumental Methods of Measurement

Polysomnography With polysomnography, it will be possible to know the stages of sleep, the total number of apneas and hypopneas, the type of apnea, the total number of micro-awakenings and the level of oxygen desaturation during sleep that, when above 4% , demonstrates important impairment during REM sleep, making patients susceptible to clinical complications.

Measurement of inspiratory muscle strength (MIP) By vacuometry In order to measure MIP, the MVD 300 digital manovacuometer (Globalmed, Porto Alegre, RS, Brazil), with a scale of 300 cmH2O, an scale increment of 1 cmH2O, and a scheduled time interval registering of at least 1 second will be used.

During the test, the patient will assume the seated position and use a nasal clip. The MIP will be measured from the residual volume (RV) until total lung capacity (CPT) is reached and three MIP measures will be performed, with a 1-min rest interval. The highest MIP values will be recorded. The values used as reference of normality, according to sex and age, will be those proposed by Neder et al (1999). After the examination, each patient's data will be digitally stored.

By POWERbreathe K-5 This electronic device aims to evaluate initial inspiratory muscle strength (S. Index) and its changes along training. Connected to a computer, it will allow graphic analysis of the measurement and data storage (LOMAX e MCCONNELL, 2009). The technical procedures to perform the measurement are the same adopted for vacuometry. There is no difference in the posture adopted, the inspiratory effort, the number of measurements performed, and the criteria of selection and acceptance of the best value. The use of this equipment will help patients to become familiarized with the inspiratory muscle training strategy that will be employed as the intervention since it is very similar to the POWERbreathe classic.

Pittsburgh Sleep Quality Scale (PSQI) The Pittsburgh Sleep Quality Scale (PSQI) is a sleep quality questionnaire that analyzes multiple sleep-related variables during the previous month. Respondents answer 19 items about themselves, of which 18 are used to calculate the score. Five additional items are completed by a bed partner or roommate, but are not used to calculate the score (Buysse et al., 1989).

The PSQI measures seven components, which evaluate subjective sleep quality (C1), sleep latency (C2), sleep duration (C3), habitual sleep efficiency (C4), sleep disturbances (C5), sleeping pills use (C6) and daytime dysfunction (C7). Scores of the subscales range from 0 to 3 and are summed to get a total score, which can range from 0 to 21. Total score greater than five suggests a significant sleep disturbance.

Berlin Snoring Questionnaire The questionnaire is composed of nine closed questions and divided into three categories (NETZER et al., 1999). Category one (01) is composed of five questions and is considered positive when two or more questions get a positive answer. Category two (02) is composed of three questions and is considered positive when two or more questions are answered positively. Category three (03) is considered positive if the individual has associated SAH or BMI ≥ 30 kg / m².

It is classified as no risk for OSAHS when the result does not present any positive category or low risk when presenting a single positive category and high risk for obstructive apnea when two or more categories are positive.

Epworth Sleepiness Scale The Epworth Sleepiness Scale (ESS) was advocated based on the observations related to the occurrence of daytime hypersomnia (HSD), through a self-administered questionnaire that evaluates the probability of falling asleep in eight situations involving daily activities.

The overall score ranges from 0 to 24, with scores above 10 suggesting the diagnosis of HSD (JOHNS, 1991).

Short Form Questionnaire - 36 (SF-36) The "Medical Outcomes Study 36-Item Short-Form Health Survey" (SF-36) is a generic questionnaire that assesses quality of life aspects that are directly related to the health of the individual. The questionnaire consists of 36 questions that assess the perception of the disease from the point of view of the patient. He evaluates eight dimensions of health: functional capacity, physical appearance, pain, general health, vitality, social aspects, emotional aspects and mental health.

Focusing on the impact of the disease on the quality of life, without focus on disease or clinical signs, becomes the great differential of this instrument. The SF-36 can be applied in several ways: patient-filled, performed by an interviewer, and even in telephone interviews.

SF-36 is a practical instrument, easy to apply, has good reliability and validity, and can be used in our population (SOÁREZ PC, 2007).

STATISTICAL ANALYSIS Data analysis will be performed by a blind investigator for the identity of the groups. The results will be expressed as mean and standard deviation for the continuous variables with Gaussian distribution, and median and internal quartiles, as an alternative. Categorical variables will be expressed as frequencies. Differences between groups will be assessed by the t student test for paired samples or by their non-parametric equivalent; between frequencies, by the chi-square test. Association between variables will be analyzed by linear regression. Values of P <0.05 will be considered significant. Statistical analysis will be performed using the statistical program SPSS, version 18.0 (Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Age equal or greater than 18 years.
* Diagnosis of obstructive sleep apnea and hypopnea syndrome (AHI> 5 events / hour).

Exclusion Criteria:

* Acute or chronic pulmonary disease, uncontrolled arterial hypertension, heart failure, chronic renal failure and neurological disease.
* Drug therapy that can influence muscle strength.
* Psychiatric illness that may make adherence to the research protocol difficult.
* Speech therapy or respiratory therapy in the last 3 months.
* Orthodontic therapy with intraoral device.
* BMI> 40 kg / m².

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index | up to 04 weeks
  measured by polysomnography

SECONDARY OUTCOMES:
Sleep quality: Pittsburgh sleep quality index | up to 04 weeks
  Assessed by the Pittsburgh sleep quality index will be measured by measuring this questionnaire at the beginning of the protocol, after 04 weeks, 08 weeks and at the end of 12 weeks.
Quality of life assessed by the The Medical Outcomes Study - Short-form 36 (SF-36) | up to 04 weeks
  assessed by the The Medical Outcomes Study - Short-form 36 (SF-36), after 04 weeks, 08 weeks and at the end of 12 weeks.
Inspiratory muscle strength | up to 04 weeks
  measured by Digital manovacuometry and Powerbreathe- K5 after 04 weeks, 08 weeks and at the end of 12 weeks.
Daytime sleepiness | up to 04 weeks
  measured by Epworth Sleepiness Scale after 04 weeks, 08 weeks and at the end of 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jocemir R Lugon, MD, PhD, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Hospital Naval Marcilio Dias, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No